CLINICAL TRIAL: NCT03730259
Title: An Innovative Tailored Intervention for Improving Children's Postoperative Recovery
Brief Title: An Innovative Tailored Intervention for Improving Children's Postoperative Recovery (WebTIPS)
Acronym: WebTIPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Zeev Kain, Professor, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1R01HD091286-01A1 [#2019-5130]; 1R01HD091286-01A1 (NIH)
Record Dates: First submitted 2018-10-15; First posted 2018-11-05 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Anxiety; Pain; Postoperative Behavior
Keywords: Pediatric; Pain; Postoperative; General Anesthesia; Anesthesia Recovery Period; Patient Satisfaction; mobile health
MeSH Terms: conditions — Anxiety Disorders; Pain; Patient Satisfaction | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WebTIPS (Experimental): A Tailored Program for Perioperative Anxiety and Pain (WebTIPS) aims at reducing perioperative anxiety and pain in children via an internet and mobile platform with short message service (SMS) two-way communication between a healthcare provider and patient/parent. The Web-based Tailored Intervention Preparation for Surgery (WebTIPS) program is developed using the conceptual framework of the Triple Aim that evaluates the intervention within the context of clinical efficacy, improved child and parent surgical experience, and reduced resource utilization during the surgical episode.
  Interventions: Other: Web-based Tailored Intervention Preparation for Surgery
- Control (No Intervention): Subjects in this attention control group, the Web-based Information (WebINFO) group will not be provided tailored content or access to two-way communication. Instead, this group will only receive basic information regarding the management of perioperative anxiety and postoperative pain via the internet and/or mobile platform.

INTERVENTIONS:
Other: Web-based Tailored Intervention Preparation for Surgery — A Tailored Internet-based Preparation Program for Perioperative Anxiety and Pain (WebTIPS) is developed using the conceptual framework of the Triple Aim that evaluates the intervention within the context of clinical efficacy, improved child and parent experience, and reduced resource utilization during the surgical episode. WebTIPS aims at reducing perioperative anxiety and pain in children via an internet-based platform with short message service (SMS) two-way communication between a healthcare provider and patient.
  Other Names: WebTIPS
  Arms: WebTIPS

SUMMARY:
The goal of this randomized trial is to examine the effectiveness of a tailored Internet-based Preparation Program (WebTIPS) in reducing anxiety and improving the recovery process in children undergoing surgery. Two hospitals and all parent-child dyads and healthcare providers (HCPs) will be randomized to either a Web-based Tailored Intervention Preparation for Surgery (WebTIPS) Group or to a Web-based Information (WebINFO) Group, the attention control group. The WebTIPS group will receive the newly developed intervention with short message service (SMS) two-way communication between an HCP and patient, while the WebINFO Group will only receive an internet and mobile platform with information on the management of preoperative anxiety and perioperative pain. The aims of this study are to:

Primary aim:

Quality of Clinical Care:

Determine whether and to what extent WebTIPS is more effective than an attention control intervention in reducing preoperative anxiety among children ages 1-12 years old undergoing anesthesia and outpatient surgery.

Secondary aims:

Quality of Clinical Care:

1. Examine the impact of WebTIPS on Post-Anesthesia care unit based postoperative clinical recovery parameters, such as pain and emergence delirium.
2. Examine the impact of WebTIPS on home-based postoperative clinical recovery parameters such as pain, new onset behavioral changes and return to normal daily activity over 2 weeks.
3. Determine if the use of WebTIPS reduces parental preoperative anxiety.

Experience of Care:

Examine the effects of WebTIPS on parental satisfaction with the overall experience of the surgical episode.

Cost of Care/Resource Use:

Determine if WebTIPS modifies healthcare resource use, as measured by 30-day charges adjusted for Medicaid cost-to-charge ratios.

DETAILED DESCRIPTION:
The proposed clustered two-arm single blind, randomized trial of two children's hospitals: CHOC Children's (CHOC) and Seattle Children's Hospital. Approximately 620 patients and their families will be recruited in total. This study will examine the effectiveness of a tailored Internet-based Preparation Program (WebTIPS) aimed at reducing anxiety and improving the recovery process in children undergoing surgery via parent and child interactive preparation modules. Each study site will have a permuted block group assignment stratified by surgical severity. Within each surgical severity group, patients and their families will be randomized to either a Web-based Tailored Intervention Preparation for Surgery (WebTIPS) Group or to a Web-based Information (WebINFO) Group, the attention control group. The WebTIPS group will receive the newly developed interactive intervention with short message service (SMS) two-way communication between a clinician and patient. Conversely, the WebINFO Group will only receive an internet and mobile platform with information on the management of preoperative anxiety and postoperative pain. Objective measures of children's preoperative anxiety and postoperative recovery will be collected prior and during the experimental period.

Patients and their parents in the intervention group will learn through the internet and mobile platforms that implementing strategies and ways to adjust behavior, such as distraction and medical reinterpretation, directs the child's attention away from their own distress or fear. This group will also have access to a SMS messaging system to allow for patient/parent-provider two-way interaction and two-way sharing of information so health care providers learn about parents' coping styles.

Child's anxiety (assessed through the modified Yale Preoperative Anxiety Scale-mYPAS) during induction will be assessed at two points, a) entering the operation room (OR) and b) introduction of the anesthesia mask to the child. If parents accompanied the child into the OR, their anxiety will be rated as they leave the OR (state-trait anxiety inventory-STAI). Also, parents answer baseline questionnaires aimed at capturing demographics (e.g. age, sex), as well as parental coping (through the Miller behavioral style scale), and child temperament (through the emotional, activity, and shyness temperament survey). In the holding area and separation, a research assistant who is blinded to group assignment will rate child anxiety (mYPAS) and ask parent anxiety (STAI), and also assess child/parent anxiety at separation to the OR (mYPAS, STAI). Postoperative analgesic consumption, behavioral and recovery measures will also be collected.

ELIGIBILITY:
Inclusion Criteria:

Children:

* Children scheduled to undergo anesthesia and outpatient surgery.
* Children whose health status is American Society of Anesthesiologists (ASA) physical status I-III will be recruited for this study.
* Only children who are in the normal range of development will be recruited for this study

Parents:

* Parents of children who are enrolled in the study.

Healthcare Providers:

* Anesthesia care providers in the two study hospitals
* Nurses who provide preoperative nursing care to children who are about to undergo surgery in the two study hospitals

Exclusion Criteria:

Children:

* Patients with health status defined by ASA status IV-V
* Children who are not in the normal range of development and who are visually impaired will be excluded from this study.
* Children with visual impairment.

Parents:

* Parents who refuse to be part of the study and whose children are not eligible for the study.
* Parents who are visually impaired.

Healthcare Providers:

* Anesthesiologists who refuse to be part of the study
* Nurses who refuse to be part of the study

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 659 (Actual)
Dates: Start 2019-04-12 (Actual); Primary Completion 2022-04-05 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Assess children's domains of behavior indicating anxiety [Activity, Emotional expressivity, State of arousal, Vocalization and Use of parents] | Day of surgery (Holding Area, Separation, Entrance to operating room, and placement of the anesthesia mask)
  Child anxiety is assessed using the Modified Yale Preoperative Anxiety Scale (mYPAS) in four time points: the holding area, separation, entrance to the operating room, and the placement of the anesthesia mask. The mYPAS is an observational measure of preoperative anxiety in children consisting of 27 items in five domains of behavior indicating anxiety in young children (Activity, Emotional expressivity, State of arousal, Vocalization and Use of parents). For each category the child is scored from 1-4 (however in vocalization it is 1-6). The mYPAS total score is a sum of all categories for all time points, and ranges from 0 to 100 with higher scores indicating greater anxiety.

SECONDARY OUTCOMES:
Change in children's postoperative pain using the Faces Pain Scale-Revised (FPS-R) | Every 15 minutes for 1-2 hours while patient is in the post-anesthesia care unit
  Nurses blinded to treatment conditions will assess children's pain through the Faces Pain Scale-Revised (FPS-R) every 15 minutes in the post-anesthesia care unit. The FPS-R is scaled from 0-10 using diagrams of cartoon faces expressing pain with scoring increments of 0, 2, 4, 6, 8, and 10, in which '0' = 'no pain' and '10' = 'very much pain.' Children are asked to pick the face and corresponding number that best describes their pain. Higher scoring increments on the scale suggest greater pain.
Assess Pediatric Anesthesia Emergence Delirium [Emergence status and Psychometric Evaluation in children] | Baseline (Post-Anesthesia Care Unit)
  Emergence status will be assessed through the Pediatric Anesthesia Emergence Delirium Scale (PAED). Items rated on a 5-point rating scale from 0 ("extremely") to 4 ("not at all"). The PAED rating scale consists of five psychometric items ("child makes eye contact with the caregiver", "child's actions are purposeful," "child is aware of the surroundings," "child is restless," "child is inconsolable") for the measurement of ED in children. Items are summed up for a total score that directly increases with the degree of emergence delirium.
Change in children's pain intensity using the Postoperative Pain Measure (PPPM) | Days 1-14 after surgery, twice a day
  Postoperative pain intensity will be assessed through the 15-item Postoperative Pain Measure (PPPM) in which parents can indicate the presence or absence of each of the 15 behavioral indicators of pain by selecting either "Yes" or "No" for each question. In this scale, "0: Yes" and "1: No." A total score is achieved by summing all 15 items--higher scores suggest greater pain intensity. The questions on this scale are specific to postoperative pain (e.g. Refuse to eat? Eat less than usual?).
Change in children's postoperative maladaptive behaviors using the Post-Hospitalization-Behavior-Questionnaire for Ambulatory Surgery | Days 5, 7, and 14 after surgery
  Parents will assess specific behaviors in the postoperative period through the Post-Hospitalization-Behavior-Questionnaire for Ambulatory Surgery (PHBQ-AS). This measure consists of 11 items and six categories of anxiety: General Anxiety, Separation Anxiety, Sleep Anxiety, Eating Disturbances, Aggression Against Authority, and Apathy/Withdrawal. This measure is scored on a 5-point Likert-type scale with responses ranging from "Much less than before" to "Much more than before."
  An average score is achieved from the items.The total PHBQ-AS score produces a continuous variable with higher values above 3 (the midpoint) indicating greater maladaptive behavioral changes, lower values below three indicating improvements in behavioral change, and values equal to 3 indicating no behavioral change.
Change in children's return to normal activity using the Pediatric Quality of Life (PedsQL) questionnaire | Days 1-14 after surgery, twice a day
  Parents are asked to report on the child's health related quality of life using the pediatric quality of life questionnaire (PedsQL). The measure incorporates a generic module and has categories of physical, emotional, social, and school functioning. Questions like, "I have trouble sleeping." are on a 5-point Likert scale from 0 ("Never") to 4 ("Almost Always").
  For this scale, the scores are transformed where "0=100, 1=75, 2=50, 3= 25, and 4=0." Higher transformed scores on the scale suggest a better health related quality of life. These responses are useful in understanding return to normal activity.
State-Trait Anxiety Inventory (STAI) (parent self-report) | Day of surgery (Holding area, separation, & Operating room)
  Only the Trait section of the questionnaire is administered to parents to assess their self-reported anxiety. Items rated on a 4-point Likert Scale from 1 ("Almost Never") to 4 ("Almost Always").Higher scores suggest higher levels of anxiety.
Assess parent satisfaction outcomes using the National Research Council (NRC) Picker satisfaction survey | Day 30 after surgery
  Given that WebTIPS changes anxiety and pain, expedites the recovery process, and provides healthcare providers with data to personalize and assist the entire surgical process,we are interested in the parent satisfaction outcomes. Parent satisfaction scores will be evaluated through the National Research Council (NRC) Picker satisfaction survey. The questions on this survey evaluate satisfaction with the most recent hospital stay (e.g. Did the providers give you enough information about each choice?). Each question presents a multiple choice response of either "Yes-definitely, Yes-somewhat, and No." For each question, positive scores transformed as a percentage will represent how many participants filled out the most satisfied response.
Change in children's postoperative pain using the Faces, Legs, Arms, Cry and Consolability pain scale (FLACC) | Every 15 minutes for 1-2 hours while patient is in the post-anesthesia care unit
  Nurses blinded to treatment conditions will assess children's pain through the Faces, Legs, Arms, Cry, and Consolability (FLACC) pain scale every 15 minutes in the post-anesthesia care unit. In each of the categories (faces, legs, arms, cry, and consolability) the behaviors are scored from 0 to 2. By summing the result of all five categories, the FLACC scale yields a total score of 0-10 with higher scores indicating greater pain.
Change in children's postoperative pain using the visual analog scale (VAS) | Every 15 minutes for 1-2 hours while patient is in the post-anesthesia care unit
  Parents will report children's postoperative pain through the visual analog scale (VAS). The VAS is presented as a sliding scale (100 mm line), and yields scores from '0: not anxious' to '100: very anxious.'
Change in children's pain intensity using the Faces Pain Scale-Revised (FPS-R) | Days 1-14 after surgery, twice a day
  Pain intensity will also be measured through the FPS-R. Parents will assess children's pain through the Faces Pain Scale-Revised (FPS-R). The FPS-R is scaled from 0-10 using diagrams of cartoon faces expressing pain with scoring increments of 0, 2, 4, 6, 8, and 10, in which '0' = 'no pain' and '10' = 'very much pain.' Children are asked to pick the face and corresponding number that best describes their pain. Higher scoring increments on the scale suggest greater pain.

OTHER OUTCOMES:
Assess children's temperament using the Emotional, Activity, Sociability, and Impulsivity temperament scale (adjusting variable) | 5 days before surgery
  The Emotional, Activity, Sociability, and Impulsivity (EASI) temperament scale will be used in order to assure the study groups are comparable.The instrument includes 20 items in four behavioral categories: Emotionality, Activity, Sociability, and Impulsivity. This parent-report scale is on 5-point Likert-type scale and the responses range from "1: A little" to "5: A lot." Items are summed, and total scores on the EASI suggest characteristics that are indicative of that behavioral category.
Assess parent behavioral coping and style using Miller Behavioral style scale (adjusting variable) | 5 days before surgery
  Through the Miller behavioral style (MBSS) scale, parents will be introduced to four scenarios of stressful situations (dentist, aeroplane, hostage, and dismissal). After, parents are prompted to select any of eight coping options that most apply to them (e.g. I would try to sleep, I would do mental puzzles in my mind). Four of the eight options represent characteristics of information seekers or monitors, while the other four options represent characteristics of avoidants or blunters. From this scale, a total monitoring, total blunting, and a summary score (total blunting minus total monitoring) are derived. Higher scores indicate higher degree of monitoring coping. Scores above the median of 4 will be categorized as "high monitors" whereas participants with scores below the median will be categorized as "low monitors." Results from this measure are indicative of parent coping style, and how well parents process and digest information.

CONTACTS AND LOCATIONS:
Overall Officials: Zeev Kain, MD, MBA, Principal Investigator — UC Irvine Medical Center, Dept. of Anesthesiology and Perioperative Care
Locations (2):
- United States (2):
  - CHOC Children's Hospital, Orange, California
  - Seattle Children's Hospital, Seattle, Washington